CLINICAL TRIAL: NCT05144945
Title: A Phase III Randomized, Modified Double-blind, Active-controlled, Multi-center Study to Describe the Immunogenicity and Safety of the Quadrivalent Recombinant Influenza Vaccine (RIV4) Versus a Quadrivalent-inactivated Influenza Vaccine (IIV4) (Fluarix® Quadrivalent) in Participants 18 Years of Age and Older in South Korea
Brief Title: Study Describing the Immunogenicity and Safety of Quadrivalent Recombinant Influenza Vaccine (RIV4) Versus a Licensed Quadrivalent-inactivated Influenza Vaccine (IIV4) (Fluarix® Quadrivalent) in Participants 18 Years of Age and Older in South Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAP00016; U1111-1253-2122 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-11-17; First posted 2021-12-06 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Influenza (Healthy Volunteers)
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; fluarix

STUDY DESIGN:
Intervention Model Description: In each age group (18-49 and >= 50 years of age), participants were randomized in a 1:1 ratio to each of the vaccines.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind: A designated unblinded administrator administered the appropriate vaccine but was not involved in the immunogenicity and safety assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) (Experimental): Participants received a single intramuscular (IM) injection of 0.5 milliliters (mL) RIV4 on Day 1.
  Interventions: Biological: Quadrivalent Recombinant Influenza Vaccine (RIV4)
- Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4) (Active Comparator): Participants received a single IM injection of 0.5 mL IIV4 on Day 1.
  Interventions: Biological: Quadrivalent inactivated influenza vaccine (IIV4)

INTERVENTIONS:
Biological: Quadrivalent Recombinant Influenza Vaccine (RIV4) — Solution for intramuscular injection
  Arms: Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4)
Biological: Quadrivalent inactivated influenza vaccine (IIV4) — Suspension for intramuscular injection
  Other Names: Fluarix®
  Arms: Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)

SUMMARY:
* To describe the immune response induced by quadrivalent recombinant influenza vaccine (RIV4) and Quadrivalent-inactivated Influenza Vaccine (IIV4) in 18-49 and greater than or equal to (>=) 50 years of age participants by hemagglutination inhibition (HAI) measurement method.
* To describe the safety profile of all participants in RIV4 and IIV4 groups.

DETAILED DESCRIPTION:
The duration of each participant's participation was approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged >=18 years on the day of inclusion.
* Participants who were overtly healthy as determined by medical evaluation including medical history, physical examination.
* Able to attend all scheduled visits and complied with all study procedures.
* Informed consent form was signed and dated.
* A female participant was eligible to participate if she was not pregnant or breastfeeding and one of the following conditions applies:

Was of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile OR Was of childbearing potential and agreed to use an effective contraceptive method or abstinence from at least 4 weeks prior to the study intervention administration until at least 4 weeks after study intervention administration.

A female participant of childbearing potential must had a negative highly sensitive pregnancy test (urine) before the first dose of study intervention.

Exclusion Criteria:

Participants were excluded from the study if any of the following criteria applied:

* Participation at the time of study enrollment, or in the 6 months preceding the study vaccination, or planned participation during the present study period in another clinical study investigating involving an Investigational Medical Product (IMP) (vaccine, drug), medical device, or medical procedure or in any other type of medical research.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the study vaccination or planned receipt of any vaccine prior to Visit 2.
* Previous vaccination against influenza (in the preceding 6 months) with either the study vaccine or another vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Known or suspected abnormal immune function: immunosuppression, suspected congenital or acquired immunodeficiency based on medical history and physical examination, or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy, or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances.
* Thrombocytopenia or bleeding disorder, contraindicating IM vaccination based on the Investigator's judgment.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction that in the opinion of the Investigator might interfere with the study conduct or completion.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion (Chronic illness may include, but is not limited to, cardiac disorders, renal disorders, auto-immune disorders, diabetes, psychiatric disorders, or chronic infection).
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >=38.0°C). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Personal or family history of Guillain-Barré syndrome.
* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that was stable at the time of vaccination in the absence of therapy and participants who had a history of neoplastic disease and had been disease-free for >= 5 years).
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse) of the Investigator or employee with direct involvement in the proposed study.

The above information was not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Investigational Site Number :4100003, Ansan-si, Gyeonggi-do
  - Investigational Site Number :4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100002, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Choi WS, Lee J, Ottaviano C, Samson S, Peng L, Shin S, Choe S, Kim WJ. Immunogenicity and safety of quadrivalent recombinant influenza vaccine in Korean adults: Phase III, randomized study. Vaccine. 2025 Aug 30;62:127521. doi: 10.1016/j.vaccine.2025.127521. Epub 2025 Aug 5. PMID 40752250
- See also: VAP00016 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25369&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 active sites in South Korea from 07 December 2021 to 01 September 2022.
Pre-assignment Details: A total of 301 participants were enrolled and randomized in the study.
Period: Overall Study
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Started | 150 | 151
Safety Analysis Set (Participants who received a dose of the study vaccine and were analyzed according to the vaccine they actually received.) | 149 | 151
Completed | 149 | 151
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4): Participants received a single IM injection of 0.5 mL RIV4 on Day 1.
- Total: Total of all reporting groups
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4) | Total
Number analyzed (Participants) | 150 | 151 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (11.9) | 46.1 (12.6) | 46.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 89 | 184
  Male | 55 | 62 | 117
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies at Day 1- Per Protocol Analysis Set (PPAS)
Description: GMTs of anti-influenza antibodies were measured using hemagglutination inhibition (HAI) assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages. Titers were expressed in terms of 1/dilution.
Time Frame: Day 1 (pre-vaccination)
Population: Analysis was performed on PPAS population that included all randomized participants who received a dose of the study vaccine and had a post-vaccination blood sample. Participants with protocol deviations were excluded from the PPAS.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 145 | 150
titers
  A/H1N1 | 30.8 [24.7 to 38.3] | 38.9 [31.7 to 47.7]
  A/H3N2 | 50.1 [40.7 to 61.7] | 47.5 [39.1 to 57.6]
  B/Victoria | 109 [86.6 to 136] | 104 [83.2 to 130]
  B/Yamagata | 237 [185 to 302] | 262 [213 to 323]

2. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies at Day 1- Full Analysis Set (FAS)
Description: GMTs of anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages. Titers were expressed in terms of 1/dilution.
Time Frame: Day 1 (pre-vaccination)
Population: Analysis was performed on FAS population that included all randomized participants who received a dose of the study vaccine and had a post-vaccination blood sample. Participants were analyzed according to the intervention to which they were randomized.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
titers
  A/H1N1 | 29.8 [24.0 to 37.1] | 38.7 [31.6 to 47.4]
  A/H3N2 | 49.3 [40.1 to 60.6] | 47.2 [38.9 to 57.2]
  B/Victoria | 104 [83.2 to 131] | 103 [81.8 to 128]
  B/Yamagata | 239 [188 to 304] | 259 [210 to 319]

3. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies at Day 29- PPAS
Description: as for outcome 2
Time Frame: Day 29 (post-vaccination)
Population: Analysis was performed on PPAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 145 | 150
titers
  A/H1N1 | 961 [784 to 1177] | 868 [732 to 1030]
  A/H3N2 | 643 [529 to 781] | 378 [321 to 445]
  B/Victoria | 646 [523 to 798] | 490 [413 to 580]
  B/Yamagata | 1268 [1072 to 1499] | 897 [782 to 1029]

4. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies at Day 29- FAS
Description: as for outcome 2
Time Frame: Day 29 (post-vaccination)
Population: Analysis was performed on FAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
titers
  A/H1N1 | 955 [783 to 1164] | 863 [728 to 1022]
  A/H3N2 | 649 [535 to 787] | 379 [323 to 446]
  B/Victoria | 640 [520 to 788] | 486 [410 to 576]
  B/Yamagata | 1268 [1076 to 1495] | 899 [784 to 1031]

5. Primary Outcome: Geometric Mean Fold-rise (GMFR) for Influenza Vaccine Antibodies-PPAS
Description: GMTs of anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages. GMFR were calculated as the ratio of GMTs post-vaccination (on Day 29) and pre-vaccination (on Day 1).
Time Frame: Day 1 (pre-vaccination) and Day 29 (post-vaccination)
Population: Analysis was performed on PPAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 145 | 150
ratio
  A/H1N1 | 31.2 [25.2 to 38.8] | 22.3 [17.9 to 27.8]
  A/H3N2 | 12.8 [10.2 to 16.1] | 7.96 [6.43 to 9.87]
  B/Victoria | 5.95 [4.82 to 7.34] | 4.70 [3.82 to 5.79]
  B/Yamagata | 5.35 [4.36 to 6.58] | 3.42 [2.85 to 4.10]

6. Primary Outcome: Geometric Mean Fold-rise (GMFR) for Influenza Vaccine Antibodies-FAS
Description: as for outcome 5
Time Frame: Day 1 (pre-vaccination) and Day 29 (post-vaccination)
Population: Analysis was performed on FAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
ratio
  A/H1N1 | 32.0 [25.8 to 39.6] | 22.3 [17.9 to 27.7]
  A/H3N2 | 13.2 [10.5 to 16.4] | 8.04 [6.49 to 9.95]
  B/Victoria | 6.14 [4.99 to 7.55] | 4.74 [3.86 to 5.83]
  B/Yamagata | 5.31 [4.33 to 6.51] | 3.47 [2.89 to 4.17]

7. Primary Outcome: Percentage of Participants Achieving Seroconversion Against Influenza Vaccine Antibodies-PPAS
Description: Anti-influenza antibodies were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages. Seroconversion was defined as either a pre-vaccination titer less than (<) 1:10 (1/dilution) and a post-vaccination titer >=1:40 (1/dilution) or a pre-vaccination titer >= 1:10 (1/dilution) and a >= four-fold increase in post-vaccination titer at Day 29.
Time Frame: Day 29 (post-vaccination)
Population: Analysis was performed on PPAS population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 145 | 150
percentage of participants
  A/H1N1: number analyzed (Participants) | 139 | 138
  A/H1N1 | 95.9 [91.2 to 98.5] | 92.0 [86.4 to 95.8]
  A/H3N2: number analyzed (Participants) | 131 | 112
  A/H3N2 | 90.3 [84.3 to 94.6] | 74.7 [66.9 to 81.4]
  B/Victoria: number analyzed (Participants) | 106 | 84
  B/Victoria | 73.1 [65.1 to 80.1] | 56.0 [47.7 to 64.1]
  B/Yamagata: number analyzed (Participants) | 100 | 71
  B/Yamagata | 69.0 [60.8 to 76.4] | 47.3 [39.1 to 55.6]

8. Primary Outcome: Percentage of Participants Achieving Seroconversion Against Influenza Vaccine Antibodies-FAS
Description: as for outcome 7
Time Frame: Day 29 (post-vaccination)
Population: Analysis was performed on FAS population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
percentage of participants
  A/H1N1: number analyzed (Participants) | 143 | 139
  A/H1N1 | 96.0 [91.4 to 98.5] | 92.1 [86.5 to 95.8]
  A/H3N2: number analyzed (Participants) | 135 | 113
  A/H3N2 | 90.6 [84.7 to 94.8] | 74.8 [67.1 to 81.5]
  B/Victoria: number analyzed (Participants) | 110 | 85
  B/Victoria | 73.8 [66.0 to 80.7] | 56.3 [48.0 to 64.3]
  B/Yamagata: number analyzed (Participants) | 101 | 72
  B/Yamagata | 67.8 [59.6 to 75.2] | 47.7 [39.5 to 56.0]

9. Primary Outcome: Percentage of Participants With Antibody Titers Greater Than or Equal to (>=) 40 (1/Dilution) Against Influenza Vaccine Antibodies-PPAS
Description: Antibody titers were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages. Percentage of participants with antibody titers >=40 (1/dilution) against influenza vaccine antibodies at Day 1 and Day 29 were reported in this outcome measure.
Time Frame: Day 1 (pre-vaccination) and Day 29 (post-vaccination)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 145 | 150
percentage of participants
  A/H1N1: Day 1: number analyzed (Participants) | 75 | 87
  A/H1N1: Day 1 | 51.7 [43.3 to 60.1] | 58.0 [49.7 to 66.0]
  A/H3N2: Day 1: number analyzed (Participants) | 101 | 98
  A/H3N2: Day 1 | 69.7 [61.5 to 77.0] | 65.3 [57.1 to 72.9]
  B/Victoria: Day 1: number analyzed (Participants) | 120 | 124
  B/Victoria: Day 1 | 82.8 [75.6 to 88.5] | 82.7 [75.6 to 88.4]
  B/Yamagata: Day 1: number analyzed (Participants) | 130 | 142
  B/Yamagata: Day 1 | 89.7 [83.5 to 94.1] | 94.7 [89.8 to 97.7]
  A/H1N1: Day 29: number analyzed (Participants) | 143 | 149
  A/H1N1: Day 29 | 98.6 [95.1 to 99.8] | 99.3 [96.3 to 100]
  A/H3N2: Day 29: number analyzed (Participants) | 144 | 149
  A/H3N2: Day 29 | 99.3 [96.2 to 100] | 99.3 [96.3 to 100]
  B/Victoria: Day 29: number analyzed (Participants) | 144 | 150
  B/Victoria: Day 29 | 99.3 [96.2 to 100] | 100 [97.6 to 100]
  B/Yamagata: Day 29 | 100 [97.5 to 100] | 100 [97.6 to 100]

10. Primary Outcome: Percentage of Participants With Antibody Titers >=40 (1/Dilution) Against Influenza Vaccine Antibodies-FAS
Description: as for outcome 9
Time Frame: Day 1 (pre-vaccination) and Day 29 (post-vaccination)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
percentage of participants
  A/H1N1: Day 1: number analyzed (Participants) | 76 | 87
  A/H1N1: Day 1 | 51.0 [42.7 to 59.3] | 57.6 [49.3 to 65.6]
  A/H3N2: Day 1: number analyzed (Participants) | 103 | 98
  A/H3N2: Day 1 | 69.1 [61.0 to 76.4] | 64.9 [56.7 to 72.5]
  B/Victoria: Day 1: number analyzed (Participants) | 122 | 124
  B/Victoria: Day 1 | 81.9 [74.7 to 87.7] | 82.1 [75.1 to 87.9]
  B/Yamagata: Day 1: number analyzed (Participants) | 134 | 143
  B/Yamagata: Day 1 | 89.9 [83.9 to 94.3] | 94.7 [89.8 to 97.7]
  A/H1N1: Day 29: number analyzed (Participants) | 147 | 150
  A/H1N1: Day 29 | 98.7 [95.2 to 99.8] | 99.3 [96.4 to 100]
  A/H3N2: Day 29: number analyzed (Participants) | 148 | 150
  A/H3N2: Day 29 | 99.3 [96.3 to 100] | 99.3 [96.4 to 100]
  B/Victoria: Day 29: number analyzed (Participants) | 148 | 151
  B/Victoria: Day 29 | 99.3 [96.3 to 100] | 100 [97.6 to 100]
  B/Yamagata: Day 29 | 100 [97.6 to 100] | 100 [97.6 to 100]

11. Primary Outcome: Percentage of Participants With Detectable Antibody Titers >= 10 (1/Dilution) Against Influenza Vaccine Antibodies- PPAS
Description: Antibody titers were measured using HAI assay for 4 influenza virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata lineages. Percentage of participants with antibody titers >=10 (1/dilution) against influenza vaccine antibodies at Day 1 and Day 29 were reported in this outcome measure.
Time Frame: Day 1 (pre-vaccination) and Day 29 (post-vaccination)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 145 | 150
percentage of participants
  A/H1N1: Day 1: number analyzed (Participants) | 119 | 135
  A/H1N1: Day 1 | 82.1 [74.8 to 87.9] | 90.0 [84.0 to 94.3]
  A/H3N2: Day 1: number analyzed (Participants) | 132 | 140
  A/H3N2: Day 1 | 91.0 [85.2 to 95.1] | 93.3 [88.1 to 96.8]
  B/Victoria: Day 1: number analyzed (Participants) | 140 | 144
  B/Victoria: Day 1 | 96.6 [92.1 to 98.9] | 96.0 [91.5 to 98.5]
  B/Yamagata: Day 1: number analyzed (Participants) | 140 | 149
  B/Yamagata: Day 1 | 96.6 [92.1 to 98.9] | 99.3 [96.3 to 100]
  A/H1N1: Day 29 | 100 [97.5 to 100] | 100 [97.6 to 100]
  A/H3N2: Day 29 | 100 [97.5 to 100] | 100 [97.6 to 100]
  B/Victoria: Day 29 | 100 [97.5 to 100] | 100 [97.6 to 100]
  B/Yamagata: Day 29 | 100 [97.5 to 100] | 100 [97.6 to 100]

12. Primary Outcome: Percentage of Participants With Detectable Antibody Titers >= 10 (1/Dilution) Against Influenza Vaccine Antibodies- FAS
Description: as for outcome 11
Time Frame: Day 1 (pre-vaccination) and Day 29 (post-vaccination)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
percentage of participants
  A/H1N1: Day 1: number analyzed (Participants) | 121 | 136
  A/H1N1: Day 1 | 81.2 [74.0 to 87.1] | 90.1 [84.1 to 94.3]
  A/H3N2: Day 1: number analyzed (Participants) | 135 | 141
  A/H3N2: Day 1 | 90.6 [84.7 to 94.8] | 93.4 [88.2 to 96.8]
  B/Victoria: Day 1: number analyzed (Participants) | 143 | 145
  B/Victoria: Day 1 | 96.0 [91.4 to 98.5] | 96.0 [91.6 to 98.5]
  B/Yamagata: Day 1: number analyzed (Participants) | 144 | 150
  B/Yamagata: Day 1 | 96.6 [92.3 to 98.9] | 99.3 [96.4 to 100]
  A/H1N1: Day 29 | 100 [97.6 to 100] | 100 [97.6 to 100]
  A/H3N2: Day 29 | 100 [97.6 to 100] | 100 [97.6 to 100]
  B/Victoria: Day 29 | 100 [97.6 to 100] | 100 [97.6 to 100]
  B/Yamagata: Day 29 | 100 [97.6 to 100] | 100 [97.6 to 100]

13. Primary Outcome: Number of Participants Reporting Immediate Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which did not had any casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report form (CRF) in terms of diagnosis and/or onset window post-vaccination. All participants were observed for 30 minutes after vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in the CRF.
Time Frame: Within 30 minutes post-vaccination
Population: Analysis was performed on safety analysis set that included participants who had received a dose of the study vaccine and were analyzed according to the vaccine they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
Participants | 0 | 0

14. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactions
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRF and considered as related to the study intervention administered. Solicited systemic reactions included fever, headache, malaise, myalgia, shivering, fatigue, nausea, and arthralgia.
Time Frame: Within 7 days post-vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
Participants
  Fever | 1 | 0
  Headache | 21 | 38
  Malaise | 50 | 49
  Myalgia | 64 | 64
  Shivering | 14 | 16
  Fatigue | 35 | 40
  Nausea | 7 | 6
  Arthralgia | 12 | 16

15. Primary Outcome: Number of Participants Reporting Solicited Injection Site Reactions
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRF and considered as related to the study intervention administered. Solicited injection site reactions included pain, erythema, swelling, induration, bruising and tenderness.
Time Frame: Within 7 days post-vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
Participants
  Pain | 77 | 83
  Erythema | 1 | 0
  Swelling | 2 | 2
  Induration | 1 | 1
  Bruising | 0 | 0
  Tenderness | 34 | 21

16. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which did not had any casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRF in terms of diagnosis and/or onset window post-vaccination.
Time Frame: From Day 1 up to 28 days post-vaccination (i.e., up to Day 29)
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
Participants | 16 | 13

17. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) And Adverse Events of Special Interest (AESI)
Description: A SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. A SAE which caused death of the participant was considered as fatal SAE. An AESIs were defined as one of scientific and medical concern specific to the Sponsor's study intervention, events for which ongoing monitoring and rapid communication by the investigator to the sponsor was done.
Time Frame: From Day 1 up to 6 months post-vaccination (i.e., up to Day 181)
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 149 | 151
Participants
  SAE | 0 | 0
  AESI | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AE data were collected from Day 1 up to 28 days post-vaccination. Solicited reaction data were collected within 7 days post-vaccination. SAEs data were collected from Day 1 up to 6 months post-vaccination (i.e., up to Day 181)
Description: Analysis was performed on safety analysis set. Solicited reaction was an expected adverse reaction (sign or symptoms) observed and reported under conditions prelisted (i.e., solicited) in CRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the CRF in terms of symptom and/or onset window post-vaccination. In AE section, solicited reaction Shivering was reported as Chills.
Arm/Group | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4)
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/151
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/151
Other Adverse Events (participants affected / at risk) | 96/149 | 100/151
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Quadrivalent Recombinant Influenza Vaccine (RIV4) (N=149) | Group 2: Quadrivalent-inactivated Influenza Vaccine (IIV4) (N=151)
Chills (General disorders) | 14 (14) | 16 (16)
Fatigue (General disorders) | 35 (35) | 40 (40)
Injection Site Pain (General disorders) | 82 (111) | 85 (104) — Pain events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Malaise (General disorders) | 50 (50) | 49 (49)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 16 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 64 (64) | 64 (64)
Headache (Nervous system disorders) | 23 (23) | 38 (38) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT05144945/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT05144945/SAP_001.pdf